CLINICAL TRIAL: NCT00677274
Title: Epidural Labor Analgesia in Different Cervical Dilation Diameter and the Risk of Cesarean Delivery
Brief Title: Epidural Analgesia in Different Cervix Diameter and the Rate of Cesarean Delivery
Acronym: EACDRCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NJFY-02028M03; NSR02970
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Labor Pain
Keywords: Epidural analgesia; Patient-controlled analgesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1 (Active Comparator): Epidural analgesia initiated at the cervix 0cm
  Interventions: Procedure: Epidural labor analgesia
- 2 (Active Comparator): Epidural analgesia initiated at the cervix 0.5cm
  Interventions: Procedure: Epidural labor analgesia
- 3 (Active Comparator): Epidural analgesia initiated at the cervix 1.0cm
  Interventions: Procedure: Epidural labor analgesia
- 4 (Active Comparator): Epidural analgesia initiated at the cervix 1.5cm
  Interventions: Procedure: Epidural labor analgesia
- 5 (Active Comparator): Epidural analgesia initiated at the cervix 2.0cm
  Interventions: Procedure: Epidural labor analgesia
- 6 (Active Comparator): Epidural analgesia initiated at the cervix 3.0cm
  Interventions: Procedure: Epidural labor analgesia
- 7 (Active Comparator): Epidural analgesia initiated at the cervix 4.0cm
  Interventions: Procedure: Epidural labor analgesia
- 8 (Active Comparator): Epidural analgesia initiated at the cervix 5.0cm
  Interventions: Procedure: Epidural labor analgesia

INTERVENTIONS:
Procedure: Epidural labor analgesia — Epidural analgesia initiated at the onset of regular uterine contraction
  Other Names: Peridural analgesia
  Arms: 1
Procedure: Epidural labor analgesia — Epidural analgesia initiated at the cervix diameter 0.5cm
  Other Names: Peridural analgesia
  Arms: 2
Procedure: Epidural labor analgesia — Epidural analgesia initiated at the cervix diameter 1.0cm
  Other Names: Peridural analgesia
  Arms: 3
Procedure: Epidural labor analgesia — Epidural analgesia initiated at the cervix diameter 1.5cm
  Other Names: Peridural analgesia
  Arms: 4
Procedure: Epidural labor analgesia — Epidural analgesia initiated at the cervix diameter 2.0cm
  Other Names: Peridural analgesia
  Arms: 5
Procedure: Epidural labor analgesia — Epidural analgesia initiated at the cervix diameter 3.0cm
  Other Names: Peridural analgesia
  Arms: 6
Procedure: Epidural labor analgesia — Epidural analgesia initiated at the cervix diameter 4.0cm
  Other Names: Peridural analgesia
  Arms: 7
Procedure: Epidural labor analgesia — Epidural analgesia initiated at the cervix diameter 5.0cm
  Other Names: Peridural analgesia
  Arms: 8

SUMMARY:
Epidural analgesia in the early stage of labor at cervix < 4.0cm was considered as a risk period for increasing the rate of cesarean delivery. The more recent studies and the investigators' previous data indicated epidural analgesia can be performed as early as the cervical dilation approximately 2.0cm. The investigators hypothesized that different cervix diameter had different rate of cesarean delivery. This trial would investigate the correlation amongst different cervical dilation and the risk of cesarean section in nulliparous women at term.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous women
2. > 18 years and < 45 years
3. Spontaneous labor
4. Analgesia request

Exclusion Criteria:

1. Allergy to opioids, a history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records
2. Participants younger than 18 years or older than 45 years
3. Those who were not willing to or could not finish the whole study at any time
4. Using or used in the past 14 days of the monoamine oxidase inhibitors
5. Alcohol addictive or narcotic dependent patients were excluded for their influence on the analgesic efficacy of the epidural analgesics;
6. Subjects with a nonvertex presentation or scheduled induction of labor
7. Cervical dilation was 5.0cm or greater before performing epidural puncture and catheterization.
8. Diagnosed diabetes mellitus and pregnancy-induced hypertension
9. Twin gestation and breech presentation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 780 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Rate of cesarean delivery | 10 min after successful vaginal delivery

SECONDARY OUTCOMES:
Rate of instrument-assisted delivery | 10 min after successful vaginal delivery
Indications of cesarean delivery | 10 min after cesarean section
Maternal Visual Analog Scale (VAS) rating of pain | 10 min prior to analgesia, at the cervix <4.0 cm, cervix 4.0-10.0 cm, cervix >10.0cm second stage of labor, 15min after vaginal delivery
Duration of analgesia | 0 min after analgesia to 15min after the disappearance of sensory block
Maternal satisfaction with analgesia | 30 min after the vaginal delivery
Maternal oral temperature | 0, 15, 30, 60, 120, 240, 480min after analgesia
Use of oxytocin after analgesia | 30 min after vaginal delivery
Maximal oxytocin dose | 30 min after vaginal delivery
Low back pain at 3 months after vaginal delivery | Three months after vaginal delivery
Breastfeeding success at 6 weeks after vaginal delivery | Six weeks after successful delivery
Neonatal one-minute Apgar scale | 1 min after baby was born
Neonatal five-minute Apgar scale | Five min after baby was born
Umbilical-cord gases analysis | 0 min after baby was born
Neonatal sepsis evaluation | 30 min after baby was born
Neonatal antibiotic treatment | 1 week after baby was born
Incidence of maternal side effects | 1 week after successful vaginal delivery

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China